CLINICAL TRIAL: NCT00646165
Title: Phase 1, Multicentre, Open-label, Dose Finding Trial of Forodesine in Patients With Relapsed B-cell Chronic Lymphocytic Leukemia
Brief Title: Trial of Forodesine in Patients With Relapsed B-cell Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor recruitment and change in development strategy
Sponsor: Mundipharma Research Limited (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX1777-110; 2007-000256-14
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: B-cell Chronic Lymphocytic Leukemia
Keywords: Leukemia, CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — forodesine

INTERVENTIONS:
Drug: Forodesine

SUMMARY:
To determine the dose and duration of treatment for the best overall response with Forodesine in relapsed B-cell chronic lymphocytic leukemia

DETAILED DESCRIPTION:
An open label, multi centre, three arm, dose finding Phase 1 trial with Forodesine as a single drug treatment in patients with relapsed CLL to establish dose and duration of treatment resulting in the best achievable response with Forodesine as a single drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed Binet Stage B or C B-CLL as defined by the National Cancer Institute (NCI) sponsored working group who have received up to 2 previous lines of treatment, one of which was fludarabine based. The two previous treatments could have included combination therapies.
* Patients must be ≥18 years of age, have a life expectancy of >6 months, and an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2. - Female patients must not be pregnant (as confirmed by negative pregnancy test for women of childbearing potential) and female and male patients must be willing to use effective contraception for the entire duration of treatment and 2 months thereafter.

Exclusion Criteria:

* Patients who have received more than 2 previous lines of treatment will be excluded from this study.
* Additional groups of patients who may not participate in the study include: patients who are pregnant and/or nursing; patients on corticosteroid treatment; patients with active infection (bacterial, viral or fungal) or severe infection (WHO 4th degree) within the last 3 months; patients with total bilirubin > 2 × ULN; patients with calculated creatinine clearance <70 mL/min; patients with seropositivity for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus; patients with any coexisting medical or psychological condition that would preclude participation in the required study procedures; patients who have participated in another clinical study <6 weeks prior to this study; or patients with a known hypersensitivity to the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To determine the dose and duration of treatment for the best achievable overall response and partial responders with forodesine in relapsed B-cell chronic lymphocytic leukemia (B-Cll)

SECONDARY OUTCOMES:
Assess safety & tolerability of forodesine in B-CLL in vitro sensitivity to forodesine & drug combinations including forodesine of peripheral lymphocytes of patients enrolled in study & to correlate these in vitro findings with clinical response

CONTACTS AND LOCATIONS:
Locations (1):
- H. Clinic I Provincial, Barcelona, Spain